CLINICAL TRIAL: NCT05586698
Title: Survey on Heart Rate Variability During Auricular Acupressure at Zero Point on the Left Ear in Healthy Volunteers: a Pilot Study
Brief Title: Heart Rate Variability During Auricular Acupressure at Zero Point on the Left Ear in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bui Pham Minh Man (Other)
Responsible Party: Sponsor-Investigator, Bui Pham Minh Man, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 675/HDDD-DHYD
Record Dates: First submitted 2022-10-11; First posted 2022-10-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Auricular Acupressure; Zero point

STUDY DESIGN:
Intervention Model Description: A single-blinded pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 57 participant received auricular acupressure at Zero point on the left ear. Heart rate, HRV, and elements of HRV will be recorded every 5 minutes.
  Interventions: Procedure: Auricular acupressure
- Group B (Experimental): 57 participant received sham acupressure at Zero point on the left ear. Heart rate, HRV, and elements of HRV will be recorded every 5 minutes.
  Interventions: Procedure: Auricular acupressure

INTERVENTIONS:
Procedure: Auricular acupressure — We conducted auricular acupressure at zero acupoints on the left ear with Vaccaria ear seed (Group A) or removed seed (Group B) in 20 minutes, with 2 times of auricular acupressure. The stimulation was performed for 30 seconds each time, with two pressure movements per second, resulting in a total of 60 pressure movements per stimulation.

SUMMARY:
Heart rate variability (HRV) is used to noninvasively assess the activity of the autonomic nervous system, in particular, its parts help to evaluate the cardiac sympathetic and parasympathetic activities. Increasing HRV may contribute to improving autonomic nervous system dysfunctions. In traditional medicine, acupuncture in the region of the vagus nerve distribution in the ear could increase parasympathetic activity and cause changes in HRV. Zero point located on the vagus nerve distribution is scientifically proven to enhance parasympathetic activity, however, the number of studies examining the effect of auricular acupressure at zero point on HRV is limited while this method is highly effective and convenient. In our study, we want to survey heart rate variability during auricular acupressure at Zero point on the left ear in healthy volunteers.

DETAILED DESCRIPTION:
Participants and Methods: A randomized controlled trial is conducted by comparing the changes in HRV and elements of HRV during the auricular acupressure process at zero point on the left ear in healthy volunteers. A total of 114 participants were randomly assigned to 2 groups by computer GraphPad software and the allocation was 1:1. Participants in the experimental group received auricular acupressure at the left zero point, while the control group received placebo auricular acupressure by removing the ear seed but keeping the sticker attached in the left zero point. The primary outcome was the change in heart rate variability during auricular acupressure at zero point on the left ear. This trial will be performed as randomized, controlled, and single- blinded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females were individuals aged between 20-29.
* Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials.
* Vital signs within normal range:

  * Pulse, and regularly heart rate, go together.
  * Resting heart rate: 60 - 100 beats/min.
  * Resting blood pressure: 90/60 mmHg to ≤ 140/90 mmHg.
  * Breathing rate: 16 ± 3 times/minute.
  * emperature: 36.6-37.50C.
  * SpO2 ≥ 95%.
* Body mass index (BMI): 18.5 - 23 kg/m2 .
* Had no history of cardiovascular disease, diabetes, or thyroid.
* Had no psychiatric stress problem during acupuncture day (confirmed by answering the DASS 21 questionnaire with stress points less than 15 points).
* Not currently participating in other intervention studies.
* Have no acupuncture experience yet.

Exclusion Criteria:

* Used stimulants such as beer, alcohol, coffee, and tobacco within 24 hours before conducting the study.
* Played sports 2 hours before the study.
* Had skin injuries in the area of auricular acupressure.
* Women during menstruation period, pregnancy, or breastfeeding.
* People using drugs affecting blood pressure and heart rate within 1 month.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Survey on heart rate variability during auricular acupressure at zero point on the left ear | During procedure
Survey on frequency-domain components LF (low-frequency range) and HF (high-frequency band) during auricular acupressure at zero point on the left ear | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Trinh DT, Nguyen NC, Tran AH, Bui MP, Vuong NL. Enhancing Vagal Tone, Modulating Heart Rate Variability with Auricular Acupressure at Point Zero: A Randomized Controlled Trial. Med Acupunct. 2024 Aug 21;36(4):203-214. doi: 10.1089/acu.2024.0001. eCollection 2024 Aug. PMID 39309627
- See also: Round R, Litscher G, Bahr F. Auricular acupuncture with laser. Evidence-Based Complementary and Alternative Medicine 2013;2013. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3710613/
- See also: Rajendra Acharya U, Paul Joseph K, Kannathal N, Lim CM, Suri JS. Heart rate variability: a review. Medical & Biological Engineering & Computing. 2006;44(12):1031-1051. — https://pubmed.ncbi.nlm.nih.gov/17111118/
- See also: Trinh D-TT, Nguyen Q-CT, Bui M-MP, Nguyen V-D, Thai K-M. Heart Rate Variability during Auricular Acupressure at Heart Point in Healthy Volunteers: A Pilot Study. Evidence-Based Complementary Alternative Medicine. 2022;2022. — https://pubmed.ncbi.nlm.nih.gov/35509626/
- See also: Arai Y-CP, Sakakima Y, Kawanishi J, et al. Auricular acupuncture at the "shenmen" and "point zero" points induced parasympathetic activation. Evidence-Based Complementary Alternative Medicine,. 2013;2013. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3687596/
- See also: He W, Wang X, Shi H, et al. Auricular acupuncture and vagal regulation. Evidence-Based Complementary Alternative Medicine. 2012;2012. — https://pubmed.ncbi.nlm.nih.gov/23304215/